CLINICAL TRIAL: NCT03594526
Title: Efficacy of a Nursing Intervention in the Process of Becoming a Mother, in First-time Mothers
Brief Title: Efficacy of a Nursing Intervention in First-time Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Carolina Vargas Porras, Nursing, PhD student in Nursing and Health, Associate Professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0418
Record Dates: First submitted 2018-07-06; First posted 2018-07-20 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Mothers; First Birth
Keywords: Nursing Care; Mothers; Research; Support

STUDY DESIGN:
Intervention Model Description: The assigment of the mothers to each group will be like that: The allocation will be generated in the Epidat 4.1 program. This will be done by blocks in groups of equal size, randomized 1: 1, control and intervention group. The generation will be given by an statistician who will not perform the intervention, nor the initial or final evaluations.
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking will be done to participant and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal support to become mother (Experimental): Maternal support to become mother: is an intervention based on the mid-range nursing theory of Ramona Mercer, whose purpose is to empower first-time mothers in their new maternal role, favoring the mother-child bond, strengthening social support and maternal self-efficacy, consists of:
  1. Four Home visits , in the first week; first month of baby life; at three months; and the fourth postpartum month.
  2. Four Educational sessions and support sessions for maternal empowerment in each home visit.
  3. Telephone follow-up: at 15 days; a month and a half; at two and a half months; and three and a half months postpartum.
  Interventions: Behavioral: Maternal support to become mother
- Control group: usual Care (Active Comparator): The participants will receive the usual education about the care of the mother during the puerperium, the care of the newborn, including breastfeeding.
  Interventions: Behavioral: Control Group: usual care

INTERVENTIONS:
Behavioral: Maternal support to become mother — "AMACOM-PRI": Apoyo Materno para Convertirse en Madre - Primerizas. Maternal support to become first-time mothers is an intervention based on the mid-range nursing theory of Ramona Mercer, whose purpose is to empower first-time mothers in their new maternal role, favoring the mother-child bond, strengthening social support and maternal self-efficacy, consists of.
  1. Four Home visits , in the first week; first month of baby life; at three months; and the fourth postpartum month.
  2. Four Educational sessions and support sessions for maternal empowerment in each home visit.
  3. Telephone follow-up: at 15 days; a month and a half; at two and a half months; and three and a half months postpartum.
  Arms: Maternal support to become mother
Behavioral: Control Group: usual care — This intervention is usual care, which consists of:
  1. care of the mother and her newborn during the puerperium
  2. Teaching about breastfeeding.
  Arms: Control group: usual Care

SUMMARY:
Experimental study will determine the efficacy of nursing intervention named Maternal support to become first-time mothers based on the theory of Ramona Mercer. Sequential explanatory design will be used. It is a mixed design with approach quantitative and qualitative in order to obtain a better approach of the phenomen. The approach quantitative will be randomized controlled clinical trial. The qualitative analysis of the content will be done according to Bardin.

DETAILED DESCRIPTION:
Taking into account the scientific literature related to studies in first-time mothers with healthy newborns, it can be concluded that the limited success of interventions that have been made suggests that the main areas of becoming a mother have not been addressed, either as part of the content or process of the interventions. This study will be conducted in 24 months. The sample size calculated will be 74 first-time mothers in total, which are allocated in two groups, intervention and control. Each group with 37 mothers.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum stage (for vaginal or for cesarean delivery)
* Mother of a healthy full term newborn.
* First-time mother.
* Self-declared support by her couple.
* Mother living in Bucaramanga metropolitan area

Exclusion Criteria:

* Multiple pregnancy.
* Mothers who cannot read or write.
* Diagnosis of postpartum depression, mental disorders, behavioral disorders.
* Mothers admitted to the intensive care unit after childbirth.
* Mothers with newborns hospitalized in the intensive care unit, intermediate care or minimal care.

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Scale name unabbreviated: "La escala de Adopción del Rol Materno (ARM) de la Doctora María del Carmen Garrido Hidalgo y la Doctora Marleny Marchán Coronado". | 4 Months
  Construct: This scale measures the process of maternal role adoption or "becoming mother" process; such process and this scale was created based in Ramona Mercer's theory. Conformation: It consists of 56 items distributed in 10 dimensions: 1)Interaction with the couple with respect to the baby, 2)baby acceptance, 3 Contact with the role of mother, 4)Stimulation of the baby, 5)Interaction with the family of origin regarding to the baby, 6 Baby care, 7)Maternal expressions of affection for the baby, 8)Well-being of the baby, 9)Concern and protection of the baby, 10)Knowledge and culture related to the baby. Scale Scores and Ranges: The instrument has a Likert scale (from 1 to 4). 1 = totally disagree and 4 = total agreement. The score are from 56 to 224. The classification score ranges are: low 56-180 points, medium 181-202 and high 203-224 points. The higher score across the scale indicate better adoption of the maternal role. The outcome of this scale is the sum of each linker-item.
Perceived Maternal Parenting Self-Efficacy (PMP S-E) by Dr. Christopher R. Barnes and Dr. Elvidina N. Adamson-Macedo: measures maternal self-efficacy. | 4 months
  _this scale measures Perceived Maternal Parenting Self-Efficacy.Conformation: This instrument was created by two psychologists from the University of Wolverhampton, Ireland. It has validity and reliability studies in Ireland and Brazil. It consists of 20 items distributed in 4 dimensions_ 1. Care tasks, 2. Behaviors raised, 3. Reading of behaviors or signals, 4. Situational beliefs. Scale Scores and Ranges_ the instrument has a Likert scale that goes from 1 to 4. There are 1 in totally disagree and 4 in total agreement. The instrument has a minimum score of 20 and a maximum score of 80. The higher the scores indicate greater (better) self-efficacy_
"Perinatal Infant Care Social Support Scale" (PICSS) by Dr. Patricia Leahy-Warren: Construct: measures social support and has been widely applied in first-time mothers. | 4 months
  Conformation: This instrument was created by a nurse from the University of College Cork, Ireland. It has validity and reliability tests in Ireland. Consisting of two subscales, the Structural Social Support subscale measures structural social support and the Functional Social Support subscale that measures functional social support. The latter is the one that is consistent with Ramona Mercer's nursing theory. The subscale Functional Social Support consists of 16 items distributed in 4 dimensions: 1) Informative Support, 2) Instrumental Support (Physical), 3) Emotional Support, 4)Valuation Support. Dimensions: Informative support (Minimum score of 7, maximum score of 28). Instrumental support (score range 7-28). Emotional support (score range 4- 16). Valuation support (score range from 4-16). The instrument has a Likert scale from 1 to 4; 1 for totally disagree and 4 for total agreement. Score range: 22-88. As higher the score, greater (better) Structural Social Support.
"Bond between parents and children of MSc Alix Nathalya Vargas Vásquez and Doctor Myriam Patricia Pardo Torres" | 4 months
  _measures the affective bond between parents and children. This instrument was created by two nurses from the National University of Colombia, Colombia. It has validity and reliability tests in Colombia and Ecuador. Conformation_ Consists of 24 items distributed in 4 dimensions_ 1. Emotional support, 2. Union - interaction, 3. Informative support, 4. Stress. Score and ranges_ the instrument has a Likert scale that goes from 0 to 5. The instrument has a minimum score_ 24 and maximum score_ 96. The low degree of affective bonding is 85 points or less

SECONDARY OUTCOMES:
Assessing the experience of motherhood: The Being a Mother Scale (BaM-13) - Spanish adaptation (by Drs. Lucy Marcela Vesga Gualdrón and Maria Mercedes Durán de Villalobos) | 4 months
  This instrument in its original English version was created by the psychologist Stephen Matthey and subsequently, based on this scale, with prior authorization, the nurses Dr. Vesga and Dr. Durán validated the Spanish scale. It is a self-report scale of 13 items. Cut point recommended is 9, which allows the classification of mothers according to the score obtained: greater than 9 is a risk of stress due to the maternal role and less than 9 is without risk of stress due to the maternal role.
Edinburgh Postnatal Depression Scale (EPDS) of Doctors J.L. Cox; JM Holden and R. Sagovsky (Spanish) | 4 months
  Construct: measures postpartum depression. This instrument was created by three doctors from the University of Keele, United Kingdom. It has been widely used in several countries and has validity and reliability tests also in Colombia. It is made up of items 10. The categories of the answers are given points of 0, 1, 2 and 3 according to the increase in the severity of the symptom. The points for questions 3, 5, 6, 7, 8, 9, 10 are noted in reverse order (for example, 3, 2, 1, 0). All points are added to give the total score. Score and range: Score range from 0 to 10. A score of 10+ shows the probability of a depression, but not its severity. Any number that is chosen other than "0" for question number 10, means that it is necessary to do additional evaluations immediately. The EPDS score is designed to assist clinical judgment, do not replace the complete clinical evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Materno Infantil San Luis, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nakamura Y, Takeishi Y, Ito N, Ito M, Atogami F, Yoshizawa T. Comfort with motherhood in late pregnancy facilitates maternal role attainment in early postpartum. Tohoku J Exp Med. 2015 Jan;235(1):53-9. doi: 10.1620/tjem.235.53. PMID 25744529
- [Result] Maehara K, Mori E, Tsuchiya M, Iwata H, Sakajo A, Ozawa H, Morita A, Maekawa T, Makaya M, Tamakoshi K. Factors affecting maternal confidence among older and younger Japanese primiparae at one month post-partum. Jpn J Nurs Sci. 2016 Oct;13(4):424-436. doi: 10.1111/jjns.12123. Epub 2016 May 11. PMID 27170452
- [Result] Gao LL, Xie W, Yang X, Chan SW. Effects of an interpersonal-psychotherapy-oriented postnatal programme for Chinese first-time mothers: a randomized controlled trial. Int J Nurs Stud. 2015 Jan;52(1):22-9. doi: 10.1016/j.ijnurstu.2014.06.006. Epub 2014 Jun 19. PMID 24994573
- [Result] Shorey S, Chan WC, Chong YS, He HG. A randomized controlled trial of the effectiveness of a postnatal psychoeducation programme on outcomes of primiparas: study protocol. J Adv Nurs. 2015 Jan;71(1):193-203. doi: 10.1111/jan.12461. Epub 2014 Jun 9. PMID 24909836
- [Result] Shorey S, Chan SW, Chong YS, He HG. Perceptions of primiparas on a postnatal psychoeducation programme: the process evaluation. Midwifery. 2015 Jan;31(1):155-63. doi: 10.1016/j.midw.2014.08.001. Epub 2014 Aug 13. PMID 25174540
- [Derived] Vargas-Porras C, Roa-Diaz ZM, Hernandez-Hincapie HG, Ferre-Grau C, de Molina-Fernandez MI. Efficacy of a multimodal nursing intervention strategy in the process of becoming a mother: A randomized controlled trial. Res Nurs Health. 2021 Jun;44(3):424-437. doi: 10.1002/nur.22123. Epub 2021 Mar 8. PMID 33682146